CLINICAL TRIAL: NCT04102007
Title: A Phase 3b, Multicenter, Interventional, Open-label Study of Adult Subjects With Moderate to Severe Plaque Psoriasis Who Have a Suboptimal Response to Secukinumab or Ixekizumab and Are Switched to Risankizumab
Brief Title: A Study of the Safety and Efficacy of Risankizumab in Adult Participants With Plaque Psoriasis Who Have Had a Suboptimal Response to Secukinumab or Ixekizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-164; 2019-000904-14 (EudraCT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis Risankizumab Secukinumab Ixekizumab Psoriasis Biologic
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Risankizumab (Other): Participants receive Risankizumab following suboptimal response to secukinumab or ixekizumab
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab is administered as a subcutaneous (SC) injection in pre-filled syringe (PFS).
  Other Names: SKYRIZI

SUMMARY:
This study will evaluate whether adult participants with moderate to severe plaque psoriasis who have been treated with secukinumab or ixekizumab for at least 6 months and are experiencing a suboptimal response may benefit from switching to risankizumab with regard to skin symptoms, quality of life symptoms and psoriasis symptoms.

Study duration will last for up to 64 weeks with risankizumab given by subcutaneous injection at Week 0, Week 4, and then every 12 weeks for 52 Weeks (With the last dose being administered at Week 40). An additional visit will occur at Week 8 for a physical exam and questionnaire collection. A final follow-up phone call will occur at Week 60.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe chronic plaque psoriasis for at least 6 months before Baseline (Week 0).
* Participant must have been on labeled secukinumab or ixekizumab treatment for at least 6 months and are experiencing suboptimal response at time of Screening and Baseline visits.
* Participant must have a Body Surface Area (BSA) 3%- <10% and Static Physician Global Assessment (sPGA) 2/3
* Participant must be eligible for continued biologic therapy as assessed by the investigator.

Exclusion Criteria:

* History of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis, psoriatic arthritis.
* Participant with active skin disease other than plaque psoriasis that could interfere with the assessment of plaque psoriasis.
* History of any documented active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix.
* History of major surgery within 12 weeks prior to Baseline or planned to be performed during the conduct of the trial as assessed by the investigator.
* Participant with exposure to risankizumab or any IL-23 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (57):
- United States (20):
  - Alliance Dermatology and MOHs /ID# 216001, Phoenix, Arizona
  - Burke Pharmaceutical Research /ID# 225023, Hot Springs, Arkansas
  - Arkansas Research Trials /ID# 225497, North Little Rock, Arkansas
  - Bakersfield Derma & Skin Cance /ID# 213480, Bakersfield, California
  - UC Davis Health /ID# 225367, Sacramento, California
  - CCD Research, PLLC /ID# 216062, Cromwell, Connecticut
  - Florida International Rsrch cr /ID# 224983, Miami, Florida
  - Advanced Medical Research /ID# 213484, Sandy Springs, Georgia
  - Arlington Dermatology /ID# 216000, Rolling Meadows, Illinois
  - Dawes Fretzin, LLC /ID# 216004, Indianapolis, Indiana
  - DermAssociates-Rockville /ID# 213837, Rockville, Maryland
  - Cleaver Dermatology /ID# 226137, Kirksville, Missouri
  - Central Dermatology, PC /ID# 213479, St Louis, Missouri
  - University Hospitals Case Medical Center /ID# 214795, Cleveland, Ohio
  - University of Pittsburgh MC /ID# 225644, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC /ID# 213836, Johnston, Rhode Island
  - Arlington Research Center, Inc /ID# 215526, Arlington, Texas
  - Bellaire Dermatology /ID# 225486, Bellaire, Texas
  - Modern Research Associates, PL /ID# 213835, Dallas, Texas
  - Menter Dermatology Res Inst /ID# 214002, Dallas, Texas
- Australia (4):
  - St George Dermatology & Skin Cancer Centre /ID# 213888, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 213889, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 213886, Carlton, Victoria
  - Fremantle Dermatology /ID# 213887, Fremantle, Western Australia
- Germany (8):
  - Universitaetsklinikum Erlangen /ID# 214228, Erlangen, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 215889, Frankfurt am Main, Hesse
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 215691, Berlin
  - Klinikum Ruhr Univ Bochum /ID# 225473, Bochum
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 214469, Lübeck
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 225472, Mahlow
  - Beldio Research GmbH /ID# 225471, Memmingen
  - Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 214506, Munich
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 213815, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 213812, Tel Aviv, Tel Aviv
  - HaEmek Medical Center /ID# 214059, Afula
  - Rabin Medical Center /ID# 213813, Petah Tikva
- Italy (6):
  - Istituto Clinico Humanitas /ID# 214749, Rozzano, Milano
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 214745, Bologna
  - Azienda Ospedaliero Universitaria di Cagliari- Presidio Ospedaliero /ID# 214748, Cagliari
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 214750, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 214751, Modena
  - AOU Universita degli Studi della Campania Luigi Vanvitelli /ID# 214752, Napoli
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol /ID# 214031, Badalona, Barcelona
  - Hospital Universitario Fundacion Alcorcon /ID# 214033, Alcorcón, Madrid
  - Hospital Parc de Salut del Mar /ID# 214034, Barcelona
  - Hospital Puerta del Mar /ID# 214428, Cadiz
  - Hospital Universitario La Paz /ID# 214341, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 214032, Valencia
- Taiwan (4):
  - Chung Shan Medical University Hospital /ID# 213634, Taichung
  - National Taiwan University Hospital /ID# 213630, Taipei
  - MacKay Memorial Hospital /ID# 213845, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 213631, Taoyuan
- United Kingdom (5):
  - Victoria Hospital /ID# 213881, Kirkcaldy, Fife
  - Russells Hall Hospital, Dudley /ID# 213878, Dudley
  - Leeds Teaching Hospitals NHS Trust /ID# 213880, Leeds
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 213877, Newcastle upon Tyne
  - Northern Care Alliance NHS Group /ID# 213873, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvieclinicaltrials.com/hcp/data-sharing/

REFERENCES:
- [Derived] Warren RB, Pavlovsky L, Costanzo A, Bukhalo M, Korman NJ, Huang YH, Kokolakis G, Pinter A, Ibrahim N, Zheng Y, Drogaris L, Stakias V, Soliman AM, Rubant S, Thaci D. Efficacy and Safety of Risankizumab in Patients with Psoriasis Showing Suboptimal Response to Secukinumab or Ixekizumab: Results from a Phase 3b, Open-Label, Single-Arm (aIMM) Study. Dermatol Ther (Heidelb). 2024 Dec;14(12):3273-3290. doi: 10.1007/s13555-024-01292-z. Epub 2024 Nov 8. PMID 39516454
- See also: Related info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Significant site non-compliance for this study was identified at one site since interim results were posted. As a result of this finding, participants enrolled in this trial site were not included in any final analysis. Adverse events or lab abnormalities were reported in 1 participant from this site. The participant was on risankizumab and had a non serious event of headache (assessed as mild), which did not lead to study drug discontinuation
Period: Overall Study
Arm/Group | Risankizumab
Started | 244
Completed | 205
Not Completed | 39
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 12
Not completed — Eligibility Violation | 5
Not completed — Lack of Efficacy | 6
Not completed — Protocol Deviation | 5
Not completed — Protocol Compliance | 1
Not completed — Withdrew Treatment | 2
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.81)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 65
  40 - 65 years | 150
  ≥ 65 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 227
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 214
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 64
  Germany | 65
  Italy | 27
  Spain | 17
  United Kingdom | 12
  Israel | 34
  Australia | 3
  Taiwan | 22

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Static Physician Global Assessment (sPGA) 0/1
Description: The sPGA is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.
Time Frame: At Week 16
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 140
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of sPGA 0/1 @ WK 16 = 57.4, 95% CI 2-sided [51.1 to 63.4] — Non-Responder Imputation incorporating multiple imputation to handle missing due to COVID-19 for proportion calculation and Wilson score method for confidence interval construction

2. Secondary Outcome: Proportion of Participants Achieving a sPGA Clear Response (sPGA 0)
Description: as for outcome 1
Time Frame: At Week 16
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 50
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of sPGA 0 @ WK 16 = 20.5, 95% CI 2-sided [15.4 to 26.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Participants Achieving a Dermatology Life Quality Index (DLQI) 0/1
Description: The DLQI is a self-administered, 10-question questionnaire covering 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and bother with psoriasis treatment). The response options range from 0, not affected at all, to 3, very much affected. This gives an overall range of 0 to 30 where lower scores mean better quality of life.
Time Frame: At Week 16
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 98
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of DLQI 0 or 1 @ WK 16 = 40.2, 95% CI 2-sided [34.2 to 46.4] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Participants Achieving a Psoriasis Symptoms Scale (PSS) 0
Description: The PSS is a 4-item patient-reported outcome (PRO) instrument that assesses the severity of psoriasis symptoms in patients with moderate to severe psoriasis (Appendix 8.2). The symptoms included are:
  pain, redness, itching and burning from psoriasis. Current symptom severity is assessed as a daily diary, using a 5-point scale ranging from 0 (none) to 4 (very severe).
Time Frame: At Week 16
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 51
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of PSS 0 @ WK 16 = 20.9, 95% CI 2-sided [16.3 to 26.4] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Proportion of Participants Achieving Static Physician Global Assessment (sPGA) 0/1
Description: as for outcome 1
Time Frame: At Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 152
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of sPGA 0/1 @ WK 52 = 62.3, 95% CI 2-sided [56.0 to 68.1] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Proportion of Participants Achieving a sPGA Clear Response (sPGA 0)
Description: as for outcome 1
Time Frame: At Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 66
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of sPGA 0 @ WK 52 = 27.1, 95% CI 2-sided [21.9 to 33.0] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Proportion of Participants Achieving a Dermatology Life Quality Index (DLQI) 0/1
Description: as for outcome 3
Time Frame: At Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 115
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of DLQI 0 or 1 @ WK 52 = 47.2, 95% CI 2-sided [41.0 to 53.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Proportion of Participants Achieving a PSS 0
Description: as for outcome 4
Time Frame: At Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Participants | 67
Statistical Analysis 1: Comparison: Risankizumab; Test type: Other — There is no statistical test for this study; Other; There is no test of hypothesis for this study; Proportion of PSS 0 @ WK 52 = 27.5, 95% CI 2-sided [22.3 to 33.4] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Time to Achieve sPGA 0/1
Description: as for outcome 1
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Days
  25th | 30 [29 to 38]
  Median | 57 [57 to 110]
  75th | 199 [134 to 282]

10. Secondary Outcome: Time to Achieve sPGA 0
Description: as for outcome 1
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) Population, which is defined as all subjects who had at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Risankizumab
Number analyzed (Participants) | 244
Days
  25th | 121 [113 to 201]
  Median | 370 [366 to NA] — If a participant never attained the endpoint, then the outcome was censored at the last visit where variable was measured
  75th | NA [NA to NA] — If a participant never attained the endpoint, then the outcome was censored at the last visit where variable was measured

ADVERSE EVENTS:
Time Frame: From Baseline Day 1 up to Week 52
Description: The Safety Analysis Set, which is defined as all subjects who received at least one dose of study drug in Study M19-164, was used for all safety analyses. In this study, the Safety Analysis Set is the same as the ITT population.
Arm/Group | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/244
Serious Adverse Events (participants affected / at risk) | 17/244
Other Adverse Events (participants affected / at risk) | 31/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=244)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
OEDEMATOUS PANCREATITIS (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
APHASIA (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PROSTATE CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=244)
NASOPHARYNGITIS (Infections and infestations) | 14 (18)
COVID-19 (Infections and infestations) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT04102007/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT04102007/SAP_002.pdf